CLINICAL TRIAL: NCT01702376
Title: A Randomized, Placebo-Controlled, Double-Blind, Four-way Crossover Study to Assess the Effect of Single Oral Doses of Retosiban on Cardiac Repolarization, With Moxifloxacin as a Positive Control in Healthy Volunteers
Brief Title: This Study Will Investigate the Effect of Single Oral Doses of Retosiban on Cardiac Repolarization, With Moxifloxacin as a Positive Control in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 113789
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Obstetric Labour, Premature
MeSH Terms: conditions — Premature Birth | interventions — GSK221149A; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Retosiban 100 mg (Experimental): Each subject will be randomized to single dose of retosiban 100 mg in one of the four treatment sequences.
  Interventions: Drug: Retosiban 100 mg
- Retosiban 800 mg (Experimental): Each subject will be randomized to single dose of retosiban 800 mg in one of the four treatment sequences
  Interventions: Drug: Retosiban 800 mg
- Placebo (Placebo Comparator): Each subject will be randomized to single dose of matching placebo in one of the four treatment sequences
  Interventions: Drug: Placebo
- Moxifloxacin 400 mg (Active Comparator): Each subject will be randomized to single dose of moxifloxacin 400 mg in one of the four treatment sequences
  Interventions: Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: Retosiban 100 mg — Subjects will be administered with single dose of one moxifloxacin placebo tablet, one 100 mg tablet of retosiban and 7 retosiban matched placebo tablets
  Arms: Retosiban 100 mg
Drug: Retosiban 800 mg — Subjects will be administered with single dose of one moxifloxacin placebo tablet and eight 100 mg tablets of retosiban
  Arms: Retosiban 800 mg
Drug: Placebo — Subjects will be administered with one moxifloxacin placebo tablet and eight retosiban matched placebo tablets
  Arms: Placebo
Drug: Moxifloxacin 400 mg — Subjects will be administered with one 400 mg moxifloxacin tablet and eight retosiban matched placebo tablets
  Arms: Moxifloxacin 400 mg

SUMMARY:
This will be a randomized, placebo-controlled, single, oral dose, four-way Williams crossover study design in healthy male and female subjects. The study consists of screening (28 days), treatment (1 day/dosing session) and follow-up (7 to 14 days) period and the total duration of study participation for each subject will be approximately 9 weeks. Each subject will participate in 4 dosing sessions separated by a minimum 7-day washout period. All subjects will receive single doses of retosiban 100 mg, (treatment A) retosiban 800 mg (Treatment B), moxifloxacin 400 mg (Treatment C) and placebo (Treatment D) in one of the four treatment sequences (ABDC, BCAD, CDBA, DACB) following a Williams design Twelve-lead ECGs and continuous Holter monitoring, clinical laboratory safety tests, vital sign measurements, physical examinations, adverse event reports, and pharmacokinetic samples will be collected throughout the study. In each study period, cardiac conduction will be measured using a 24-hour continuous 12-lead Holter monitor from the morning of Day 1 (dosing) until the morning of Day 2.

ELIGIBILITY:
Inclusion Criteria:

* - Male or female between 18 and 45 years of age inclusive, at the time of signing the informed consent
* A female subject is eligible to participate if she is of: child-bearing potential and agrees to use the contraception methods from time of consent until until 48 hours post last dose; Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 to 4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GlaxoSmithKline (GSK) Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight (greater than or equal to) >=50 kg and body mass index (BMI) within the range 19 to 29.9 kg/m^2
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* No significant abnormality on 12-lead ECG at screening, including the following specific requirements: ventricular rate >=40 beats per minute, PR interval less than or equal to (<=) 210 miliseconds (msec), Q waves less than (<)30 msec, QRS interval to be >=60 msec and <120 msec; the waveforms must enable the QT interval to be clearly defined; QTcB or QTcF interval must be <450 msec
* ALT, alkaline phosphatase and bilirubin <=1.5xULN (isolated bilirubin greater than (>) 1.5x upper limit of normal (ULN) is acceptable if bilirubin is fractionated and direct bilirubin <35%)

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A supine blood pressure that is persistently higher than 140/90 millimeters of mercury (mmHg).
* A supine mean heart rate outside the range 40 to 90 beats per minute (bpm).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml [milliliters]) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 ml within a 56 day period.
* Pregnant females as determined by positive serum human chorionic gonadotropin (hCG) test at screening or prior to dosing. Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* History or presence of any medically significant disease, or any disorder that would introduce additional risk or interfere with the study procedures or outcome. In particular, a family history of QT prolongation, of early or sudden cardiac death or of early cardiovascular disease.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements from 14 days before screening until the follow-up visit unless in the opinion of the Investigator and sponsor the medication will not interfere with the study or compromise subject safety.
* Serum calcium, magnesium or potassium levels outside the reference range
* History of sensitivity to quinolone antibiotics or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-10-03 (Actual); Primary Completion 2013-01-14 (Actual); Study Completion 2013-01-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QT duration corrected for heart rate by Fridericia's formula (QTcF) interval at each timepoint for retosiban as compared with time-matched placebo | Baseline (Day 1-pre-dose) and 1 hour [hr], 8 hrs, 12 hrs , 24 hrs (Day 2) post-dose and Day 7 per dosing session.
  Single 12-lead electrocardiograms (ECG)s will be obtained at each timepoint during the study using an ECG machine that automatically calculates corrected QT interval (QTc) interval. An average of at least 3 12-lead Holter ECG replicates per time point. Change = 12-lead ECG reading at each timepoint minus the baseline 12-lead ECG reading.

SECONDARY OUTCOMES:
Change from baseline in QTcF, QT duration corrected for heart rate by Bazett's formula (QTcB), and QT interval corrected for heart rate (QTci) /QTciL interval at each timepoint for 100 mg and 800 mg retosiban as compared with time-matched placebo | Baseline (Day 1-pre-dose) and 1 hour [hr], 8 hrs, 12 hrs , 24 hrs (Day 2) post-dose and Day 7 per dosing session.
  Single 12-lead ECGs will be obtained for subjects receiving 100 mg and 800 mg retosiban at each timepoint during the study using an ECG machine that automatically calculates QTc interval. An average of at least 3 12-lead Holter ECG replicates per time point. Change = 12-lead ECG reading at each timepoint minus the baseline 12-lead ECG reading
Change from baseline in QTcF, QTcB, and QTci/QTciL interval at each timepoint for moxifloxacin as compared with time-matched placebo | Baseline (Day 1-pre-dose) and 1 hour [hr], 8 hrs, 12 hrs , 24 hrs (Day 2) post-dose and Day 7 per dosing session.
  Single 12-lead ECGs will be obtained for subjects receiving moxifloxacin at each timepoint during the study using an ECG machine that automatically calculates QTc interval. An average of at least 3 12-lead Holter ECG replicates per time point. Change = 12-lead ECG reading at each timepoint minus the baseline 12-lead ECG reading.
Plasma concentrations of retosiban and GSK2847065 | Day 1 (pre-dose), 0.25 hr, 0.5 hr, 0.75 hr, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 18 hr post-dose and Day 2 per dosing session.
  Pharmacokinetic data will include plasma concentration of retosiban and GSK2847065
Maximum observed concentration (Cmax) for retosiban and GSK2847065 | Day 1 (pre-dose, 0.25 hr, 0.5 hr, 0.75 hr, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 18 hr post-dose) and Day 2 per dosing session
  Pharmacokinetic data will include Cmax of retosiban and GSK2847065
Time to maximum concentration (tmax) for retosiban and GSK2847065 | Day 1 (pre-dose, 0.25 hr, 0.5 hr, 0.75 hr, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 18 hr post-dose) and Day 2 per dosing session
  Pharmacokinetic data will include tmax of retosiban and GSK2847065
Area under the concentration-time curve over the dosing interval (AUC(0-τ)) for retosiban and GSK2847065 | Day 1 (pre-dose, 0.25 hr, 0.5 hr, 0.75 hr, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 18 hr post-dose) and Day 2 per dosing session
  Pharmacokinetic data will include AUC0-τ of retosiban and GSK2847065
Maximal change from baseline for QTcF and QTcB | Baseline (Day 1-pre-dose) and 1 hour [hr], 8 hrs, 12 hrs , 24 hrs (Day 2) post-dose and Day 7 per dosing session
  Single 12-lead ECGs will be obtained using an ECG machine that automatically calculates QTc interval. An average of at least 3 12-lead Holter ECG replicates per time point. Maximal Change from baseline = maximum 12-lead ECG reading at each timepoint minus the baseline 12-lead ECG reading
Change from baseline for other cardiac electrophysiological parameters: QT, QRS, RR, PR and ventricular rate at each timepoint | Baseline (Day 1-pre-dose) and 1 hour [hr], 8 hrs, 12 hrs , 24 hrs (Day 2) post-dose and Day 7 per dosing session
  Single 12-lead ECG will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and QTc intervals. Change from baseline for other cardiac electrophysiological will be calculated as: other cardiac electrophysiological parameters at each timepoint minus baseline value
Safety and tolerability of retosiban as assessed by change from baseline in 12-lead ECGs | Day 1 (pre-dose, 1 hr, 8 hr, 12 hr post-dose), Day 2 and Day 7
  Single 12-lead ECG will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and QTc intervals
Safety and tolerability of retosiban as assessed by change from baseline in systolic and diastolic blood pressure | Day 1 (pre-dose, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 18 hr post-dose), Day 2 and Day 7
  Vital sign measurements will be done in supine position and will include systolic and diastolic blood pressure
Safety and tolerability of retosiban as assessed by change from baseline in pulse rate | Day 1 (pre-dose, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 18 hr post-dose), Day 2 and Day 7
  Vital sign measurements will be done in supine position and will include pulse rate.
Safety and tolerability of retosiban as assessed number of adverse events | 9 weeks
  Safety and tolerability parameters will include recording of AEs, throughout the study
Safety and tolerability of retosiban as assessed by change from baseline in clinical laboratory tests | Day -1 and Day 2 and Day 7
  Clinical laboratory assessments will include hematology, clinical chemistry, routine urinalysis and additional parameters

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Stier B, Fossler M, Liu F, Caltabiano S. Effect of Retosiban on Cardiac Repolarization in a Randomized, Placebo- and Positive-controlled, Crossover Thorough QT/QTc Study in Healthy Men and Women. Clin Ther. 2015 Jul 1;37(7):1541-54. doi: 10.1016/j.clinthera.2015.05.007. Epub 2015 Jun 29. PMID 26138866
- See also: Results for study 113789 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/113789?search=study&search_terms=113789#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113789 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register